CLINICAL TRIAL: NCT03255148
Title: Influence of Oxytocin on Resting State Neurophysiological Measures
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Research Foundation Flanders (Other)
Responsible Party: Principal Investigator, Kaat Alaerts, Prof. Dr. Kaat Alaerts, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: SingleOT_REST_S56327
Record Dates: First submitted 2017-08-11; First posted 2017-08-21 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Oxytocin
Keywords: resting state; EEG; skin conductance; heart rate; oxytocin
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxytocin (Experimental): Syntocinon nasal spray (40 IU/ml; oxytocin, product code RVG 03716); single intranasal dose of 24 international units (IU; 3 puffs of 4 IU per nostril)
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): saline natriumchloride solution nasal spray; single intranasal dose (3 puffs per nostril)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — Syntocinon nasal spray
  Other Names: syntocinon
  Arms: Oxytocin
Drug: Placebo — Placebo nasal spray
  Arms: Placebo

SUMMARY:
In this study, the investigators will explore the influence of oxytocin administration on several neurophysiological responses (EEG, skin conductance and heart rate) during rest.

DETAILED DESCRIPTION:
Oxytocin is known to influence several neurophysiological measures, such as heart rate, EEG and skin conductance during specific tasks (e.g., emotion recognition, fear learning and extinction). However, not much is known about the influence of oxytocin on those measures during rest. Therefore, in this randomized, placebo controlled, double blinded study, the investigators will investigate the influence of oxytocin during a resting period of 5 minutes. Heart rate, skin conductance, respiration and EEG will be measured before and after oxytocin or placebo administration. The investigators expect that oxytocin will increase the heart rate variability and decrease the skin conductance levels. Exploratory, the investigators will conduct a cross-frequency analysis of band power and asses the relationship between distinct indexes of sympathetic / parasympathetic balance.

Please note that this study is part of a larger study in which the investigators also asses the influence of oxytocin on neurophysiological responses elicited by direct gaze

ELIGIBILITY:
Inclusion Criteria:

* right-handed
* male
* age between 18 and 35
* Normal or adjusted-to-normal vision (with lenses only)
* Dutch as mother tongue

Exclusion Criteria:

* not right-handed
* female
* age below 18 or above 35
* Need to wear glasses
* Dutch not as mother tongue

Ages: 18 Years to 38 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2018-05-18 (Actual); Study Completion 2018-05-18 (Actual)

PRIMARY OUTCOMES:
Change in heart rate variability after oxytocin administration | Assessment over 5 minutes, before and after oxytocin or placebo administration
  The influence of oxytocin administration on heart rate variability

SECONDARY OUTCOMES:
Change in skin conductance level after oxytocin administration | Assessment over 5 minutes, before and after oxytocin or placebo administration
  The influence of oxytocin administration on skin conductance level

CONTACTS AND LOCATIONS:
Overall Officials: Kaat Alaerts, PhD, Principal Investigator — KU Leuven
Locations (1):
- KU Leuven, Leuven, Belgium